CLINICAL TRIAL: NCT00871936
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety and Efficacy of SLx-4090 in Combination With Metformin in Subjects With Type 2 Diabetes
Brief Title: A Comparison of SLx-4090 in Combination With Metformin Versus Metformin Therapy Alone in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Response Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLx-4090-09-07
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 6-(4'-trifluoromethyl-6-methoxybiphenyl-2-ylcarboxamido)-1,2,3,4-tetrahydroisoquinoline-2-carboxylic acid phenyl ester; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): SLx-4090 in combination with Metformin
  Interventions: Drug: SLx-4090; Drug: Metformin
- 2 (Other): Placebo
  Interventions: Other: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: SLx-4090 — SLx-4090
  Arms: 1
Other: Placebo — matching tablets
  Arms: 2
Drug: Metformin

SUMMARY:
The purpose of this study is to determine whether SLx-4090 in combination with metformin therapy will reduce HbA1c in patients with Type 2 Diabetes more effectively than metformin therapy alone.

DETAILED DESCRIPTION:
1. HbA1c after 12 weeks
2. FPG after 12 weeks
3. Safety and tolerability
4. Plasma levels of SLx-4090

ELIGIBILITY:
Inclusion Criteria:

* HbA1c 7-11%
* On a stable dose of metformin for at least 6 weeks

Exclusion Criteria:

* Type 1 Diabetes
* Antidiabetic medication other than or in addition to metformin
* FPG > 270 mg/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Reduction in HbA1c | 12 weeks

SECONDARY OUTCOMES:
Adverse Events | 12 weeks

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Anaheim, California
  - Burbank, California
  - Los Angeles, California
  - West Palm Beach, Florida
  - Addison, Illinois
  - Auburn, Maine
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Winston-Salem, North Carolina
  - Greenville, South Carolina
  - San Antonio, Texas